CLINICAL TRIAL: NCT07280520
Title: Evaluating the Role of Luteolin Supplementation in Cellular Metabolism of Myocytes and Fat Cells by Regulating the Gene Expression of MEF2 and SREBP-1 Proteins, and Examining Its Effects on Physical Performance and Body Composition in Jordanian Athletes.
Brief Title: The Role of Luteolin Supplementation in Cellular Metabolism of Myocytes and Fat Cells, Physical Performance, and Body Composition in Athletes.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hadeel Ali Ghazzawi, Prof., University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 346 / 2025; 2025-148/2024 (Other Grant/Funding Number: University of Jordan)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Athletes
Keywords: luteolin; athlete; MEF-2; SREBP-1; anaerobic performance; body composition
MeSH Terms: interventions — Luteolin

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luteolin Supplement (Experimental): Participants in this arm receive a daily 100 mg capsule of Luteolin for 12 continuous weeks. This arm aims to evaluate the effect of the active substance on MEF2 and SREBP-1gene expression, physical performance, and body composition.
  Interventions: Dietary Supplement: luteolin
- Placebo Control (Placebo Comparator): Participants in this arm receive an identical-looking capsule containing only microcrystalline cellulose (a neutral substance) daily for 12 continuous weeks. This serves as the control against which the Luteolin group's outcomes will be compared.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: luteolin — 100 mg Luteolin (Active Ingredient), taken orally once daily for 12 weeks.
  Arms: Luteolin Supplement
Other: Placebo — Microcrystalline cellulose (Placebo), taken orally once daily for 12 weeks. The capsule is matched in size, color, and taste to the active Luteolin supplement.
  Arms: Placebo Control

SUMMARY:
A clinical trial is to determine whether Luteolin supplementation can enhance cellular metabolism and improve physical performance in apparently healthy Jordanian male athletes aged 18-35 with continuous training experience.

The main questions it aims to answer are:

* Does 12 weeks of Luteolin supplementation increase the gene expression of MEF2 (a factor promoting muscle development and endurance)?
* Does 12 weeks of Luteolin supplementation decrease the gene expression of SREBP-1 (a factor regulating fat storage)?
* Does Luteolin supplementation lead to improvements in key performance metrics, such as maximal oxygen consumption VO2 max) and anaerobic power?
* Does Luteolin supplementation positively impact body composition, specifically by reducing fat mass and increasing lean muscle mass? Researchers will compare the group receiving the active Luteolin supplement (100 mg daily) to a placebo group receiving a microcrystalline cellulose supplement (a neutral substance) to determine whether the active supplement has the desired effects on metabolism, performance, and body composition.

Participants will:

* Take one capsule (either Luteolin or placebo) daily for 12 weeks.
* Continue their usual diet and exercise regimen but restrict intake of high-Luteolin foods during the study period.
* Provide a blood sample for gene expression analysis before and after the 12-week intervention.
* Undergo performance assessments, VO2 max and Wingate test, and body composition analysis (BIA) before and after the 12-week intervention.

DETAILED DESCRIPTION:
This study is designed to evaluate Luteolin's potential to optimize metabolic health and physical performance in athletes by modulating specific transcription factors.

* Rationale: Effective management of lipid metabolism and enhanced muscle function are critical for athletic performance. Luteolin has shown in recent studies the potential to modulate gene expression, specifically activating MEF2 and downregulating SREBP-1.
* MEF2 Focus: Activation of MEF2 is linked to enhanced oxidative capacity, promotion of mitochondrial biogenesis, and improved muscle endurance, which are highly beneficial for athletes. Luteolin is thought to enhance MEF2 activity by promoting histone deacetylation.
* SREBP-1 Focus: SREBP-1 controls the expression of genes responsible for the synthesis of fatty acids and triglycerides. Downregulation of SREBP-1 is desirable for athletes to prevent excessive lipid accumulation and support better metabolic health and performance. Luteolin can inhibit the maturation of SREBP-1, reducing its activity and the expression of lipogenic genes.
* Design: A multi-center, double-blinded, placebo-controlled clinical trial will be conducted, requiring a total sample size of 50 male athletes. Outcome assessments include Real-Time PCR on blood samples for gene expression , Wingate and Vmax tests for performance , and Bioelectrical Impedance Analysis (BIA) for body composition.

ELIGIBILITY:
Inclusion Criteria:

* Gender and Age: Male volunteers aged 18 to 35 years old.

Athletic Status: Currently training male athletes with continuous sports training experience in any field (e.g., endurance, team sports, strength training).

Health Status: Apparently healthy, with no known chronic diseases or metabolic disorders that could interfere with lipid or muscle metabolism (e.g., diabetes, liver disease, kidney disease, cardiovascular disease).

Geographic Location: Must be residing in Jordan for the duration of the study and able to attend all scheduled assessment sessions at the specified study centers (University of Jordan).

Informed Consent: Must provide voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Pre-existing Conditions: Diagnosis of any chronic diseases, including cardiovascular disease, hypertension, diabetes mellitus, kidney disease, or any diagnosed neurological or immune system disorders.
* Medication Use: Currently using any prescription medications that could influence lipid metabolism, inflammatory status, or exercise performance (e.g., corticosteroids, statins, certain anti-inflammatory drugs).
* Supplement Use: Current or recent use (within the last 3 months) of any nutritional supplements Luteolin containing supplements. Failure to agree to restrict consumption of Luteolin-rich foods throughout the 12-week intervention period.
* Study Commitment: Inability or unwillingness to comply with the study protocol, including the 12-week daily capsule intake and attendance at all assessment visits.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male volunteers
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in SREBP-1 Gene Expression | Baseline (Week 0) and End of Intervention (Week 12)
  Gene expression of SREBP-1 (Sterol Regulatory Element-Binding Protein 1) measured using Real-Time Polymerase Chain Reaction (RT-PCR) on collected salivary samples. The outcome is the fold change in expression from baseline to Week 12.
Change in MEF2 Gene Expression | Baseline (Week 0) and End of Intervention (Week 12)
  Gene expression of MEF2 (Myocyte Enhancer Factor 2) measured using Real-Time Polymerase Chain Reaction (RT-PCR) on collected blood samples. The outcome is the fold change in expression from baseline to Week 12.

SECONDARY OUTCOMES:
Change in Maximal Oxygen Consumption (Vo2 max) | Baseline (Week 0) and End of Intervention (Week 12)
  VO2 max will be assessed via an incremental exercise test (e.g., Bruce protocol or similar) to measure cardiorespiratory fitness.
Change in Anaerobic Power (Wingate Test) | Baseline (Week 0) and End of Intervention (Week 12)
  Peak and average anaerobic power will be determined using the standard 30-second Wingate Anaerobic Power Test.
Change in Body Composition (Fat Mass and Lean Mass) | Baseline (Week 0) and End of Intervention (Week 12)
  Percentage of body fat and total lean muscle mass will be assessed using Bioelectrical Impedance Analysis (BIA).

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel A Ghazzawi, professor, Principal Investigator — The University of Jordan School of Agriculture
Locations (1):
- University of Jordan (UJ), Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Time Frame: Immediately following publication
Access Criteria: Data will be available upon request to researchers who provide a methodologically sound proposal and who have obtained ethical approval from a relevant Institutional Review Board (IRB) or Ethics Committee.